CLINICAL TRIAL: NCT00182208
Title: Evaluation of a Venous-Return Assist Device (Venowave) to Treat Post-Thrombotic Syndrome: A Randomized Controlled Trial
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hamilton Health Sciences Corporation (Other)
Collaborators: Health Canada (Other Government)
Organization: McMaster University (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CTMG-2005-VENOPTS; Health Canada No.:64844
Record Dates: First submitted 2005-09-12; First posted 2005-09-16 (Estimated); Last update posted 2008-07-22 (Estimated); Status verified 2008-07

CONDITIONS: Postphlebitic Syndrome
Keywords: PTS; Post phlebitic Syndrome; Activities of Daily Living; Quality of Life
MeSH Terms: conditions — Postphlebitic Syndrome; Postthrombotic Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: Veno-device (Venowave)

SUMMARY:
The purpose of this study is to determine whether daily use of a lower limb venous-return assist device, "Venowave', improves leg symptoms, ability to perform activities of daily living, and quality of life in subjects with severe PTS.

DETAILED DESCRIPTION:
Eligible consenting patients will be randomly allocated to receive either the veno-device (active or placebo for 8 weeks and crossed over for a further 8 weeks (active or placebo) following a 4 week 'wash out' period.( A randomized controlled 'crossover' study}

ELIGIBILITY:
Inclusion Criteria:

* Past History of objectively documented deep vein thrombosis
* Daily leg swelling with discomfort (i.e. report at least one of the following symptoms: heavy legs, aching legs and/or throbbing) for a minimum of 6 months
* Over 18 years of age (and of either gender).
* Villalta score of greater than 14(i.e.severe post phlebitic syndrome)

Exclusion Criteria:

* Episode of objectively documented deep vein thrombosis occurred less than 6 months before recruitment
* Subjects report that their symptoms have been unstable (worsening, improving or variable over the previous month).
* Active venous ulceration
* Baseline leg circumference greater than 50 cm (cuff will not fit subject)
* Symptomatic peripheral arterial disease Peripheral neuropathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32
Dates: Start 2004-05; Primary Completion 2005-06 (Actual); Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
Clinical Success measured with the Global Rating Instrument

SECONDARY OUTCOMES:
PTS-CCS questionnaire
Villalta Scale
Veines Quality of Life Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Martin O'Donnell, MB MRCPI, Principal Investigator — Hamilton Health Sciences Corporation; Susan R Kahn, MD FRCPC, Principal Investigator — Department of Medicine McGill University
Locations (2):
- Canada (2):
  - Henderson Research Centre, Hamilton, Ontario
  - Sir Mortimer B. Davis Jewish General Hospital, Montreal, Quebec